CLINICAL TRIAL: NCT06762431
Title: Phase I/II Open-label Study Evaluating The Safety And Efficacy of Concomitant Administration of Anti-CD19 CAR T-cell Therapy and Lenalidomide in Refractory/Relapsed Chronic Lymphocytic Leukemia Patients.
Acronym: VTB-CLL002
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vitebsk Regional Clinical Cancer Centre (Other)
Collaborators: Republican Scientific and Practical Center for children's Oncology, Hematology and Immunology (Unknown)
Responsible Party: Principal Investigator, Mikalai Katsin, Chief of Hematology/Oncology department, Vitebsk Regional Clinical Cancer Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTB-CLL002
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Chronic Lymphocytic Leukaemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: anti-CD19 CAR T-cells; Lenalidomide; Ibrutinib
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose antiCD19 CAR T-cells plus low dose Lenalidomide (Experimental): Phase 1: Determine safety of IL-7/IL-15 expanded 50x10^6 antiCD19 CAR-T cells with concomitant low dose Lenalidomide in patients with relapsed/refractory CLL. Patients will be enrolled in 3+3 fashion.
  Phase 1b: Six to nine patient expansion cohorts. If six patients are enrolled in Phase 1 then only six additional patients will be added. If three patients are enrolled in Phase 1 then nine additional patients will be treated for a total of 12 patients.
  Interventions: Drug: Lenalidomide
- Low dose antiCD19 CAR T-cell therapy plus high dose Lenalidomide (Experimental): Phase 1: Determine safety of IL-7/IL-15 expanded 50x10^6 antiCD19 CAR-T cells with concomitant high dose Lenalidomide in patients with relapsed/refractory CLL. Patients will be enrolled in 3+3 fashion. Phase 1b: Six to nine patient expansion cohorts. If six patients are enrolled in Phase 1 then only six additional patients will be added. If three patients are enrolled in Phase 1 then nine additional patients will be treated for a total of 12.
  Interventions: Drug: Lenalidomide
- High dose antiCD19 CAR T-cell therapy plus low dose Lenalidomide (Experimental): Phase 1: Determine safety of IL-7/IL-15 expanded 150x10^6 antiCD19 CAR-T cells with concomitant low dose Lenalidomide in patients with relapsed/refractory CLL. Patients will be enrolled in 3+3 fashion. Phase 1b: Six to nine patient expansion cohorts. If six patients are enrolled in Phase 1 then only six additional patients will be added. If three patients are enrolled in Phase 1 then nine additional patients will be treated for a total of 12.
  Interventions: Drug: Lenalidomide
- High dose antiCD19 CAR T-cell therapy plus high dose Lenalidomide (Experimental): Phase 1: Determine safety of IL-7/IL-15 expanded 150x10^6 antiCD19 CAR-T cells with concomitant high dose Lenalidomide in patients with relapsed/refractory CLL. Patients will be enrolled in 3+3 fashion. Phase 1b: Six to nine patient expansion cohorts. If six patients are enrolled in Phase 1 then only six additional patients will be added. If three patients are enrolled in Phase 1 then nine additional patients will be treated for a total of 12.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Dose Level 1
  Other Names: Revlimid
  Arms: High dose antiCD19 CAR T-cell therapy plus low dose Lenalidomide; Low dose antiCD19 CAR T-cells plus low dose Lenalidomide
Drug: Lenalidomide — Dose Level 2
  Other Names: Revlimid
  Arms: High dose antiCD19 CAR T-cell therapy plus high dose Lenalidomide; Low dose antiCD19 CAR T-cell therapy plus high dose Lenalidomide

SUMMARY:
This is a Phase I/II interventional, open-label treatment study designed to evaluate the safety and efficacy of concomitant therapy with anti-CD19 CAR T-cells and Lenalidomide in adult patients with relapsed/refractory chronic lymphocytic leukemia (CLL) who have been pretreated with Ibrutinib for 3 months prior to leukapheresis.

DETAILED DESCRIPTION:
This is a single-center, open-label study. After meeting the eligibility criteria and enrolling in the trial, patients will take Ibrutinib for 3 months up to Day -1. Leukapheresis for the collection of autologous lymphocytes will take place 2-3 weeks before Day 0. Once the cells have been manufactured, patients will proceed to lymphodepleting chemotherapy with cyclophosphamide and fludarabine from Days -5 to -3, followed by the infusion of anti-CD19-4-1BB-CD3z CAR T-cells at two fixed dose levels: DL1 (50 x 10^6 cells) and DL2 (150 x 10^6 cells), concomitantly with Lenalidomide intake. Lenalidomide maintenance at the dose of 25 mg will be administered from Day +30 for 3 months.

The main purposes of the Phase I part are:

* To preliminarily explore the safety (incidence of CRS, ICANS, HLH, infections, late ICAHT, and cytopenias) and tolerability.
* To explore the pharmacokinetics of CAR-T cells.

The main purposes of the Phase II part are:

* Overall response rate, including complete response (CR) and partial response (PR) rates.
* Duration of response (DOR).
* Progression-free survival rates.
* Overall survival rates.
* MRD negativity rates measured by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Documented CD19+ CLL or SLL
* Patients must have failed at least 1 prior regimen
* Patients must be currently receiving ibrutinib for at least 3 months prior to enrollment in the study and:
* Not experiencing any ≥ grade 2 non-hematologic ibrutinib-related toxicity
* ECOG Performance status 0 or 1
* 18 years of age and older
* Adequate organ system function including:

Creatinine < 1.6 mg/dl ALT/AST < 3x upper limit of normal Total Bilirubin <2.0 mg/dl with the exception of patients with Gilbert syndrome; patients with Gilbert syndrome may be included if their total bilirubin is ≥ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN.

* Have no active GVHD and require no immunosuppression
* Are more than 6 months from transplant
* No contraindications for leukapheresis
* Left Ventricular Ejection fraction >50%
* Gives informed consent

Exclusion Criteria:

* CLL patients with known or suspected transformed disease (i.e. Richter's transformation).
* Pregnant or lactating women.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications.
* Any uncontrolled active medical disorder
* HIV infection.
* Patients with active CNS involvement with malignancy.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification.
* Subjects with clinically apparent arrhythmia or arrhythmias who are not stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events incidence | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology/Oncology department, Vitebsk, Select A State, Belarus

IPD SHARING:
Plan to Share IPD: Undecided